CLINICAL TRIAL: NCT03233971
Title: Patients' and Caregivers' Attitudes Towards Deprescribing in the Asian Community Setting
Brief Title: How do Older Adults and Caregivers Feel About Their Medications?
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Collaborators: Guardian (Unknown); NTUC Unity (Unknown); Watsons (Unknown); Kwong Wai Shiu Hospital (Unknown); Ang Mo Kio - Thye Hua Kwan Hospital (Other); Khoo Teck Puat Hospital (Other); National University Hospital, Singapore (Other); Singapore General Hospital (Other); Tan Tock Seng Hospital (Other); National Healthcare Group Pharmacy (Unknown)
Responsible Party: Principal Investigator, Kua Chong Han, Principal Investigator, Monash University
Other Study IDs: 2017-8872
Record Dates: First submitted 2017-07-24; First posted 2017-07-31 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Deprescribing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults
  Interventions: Other: rPATD Questionnaire
- Caregivers
  Interventions: Other: rPATD Questionnaire

INTERVENTIONS:
Other: rPATD Questionnaire — A 5-point Likert scale questionnaire consisting of 22 questions for older adults, and 19 questions of caregivers.

SUMMARY:
The aim of this study is to study patients' and caregivers' perspectives towards deprescribing using the Revised Patients' Attitudes Towards Deprescribing (rPATD) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Older adults' inclusion criteria:

  * age at least 65 years;
  * taking one or more long-term prescription medication;
  * have not participated in this anonymous questionnaire previously
* Caregivers' inclusion criteria:

  * currently an informal caregiver for an older adult (defined as having any role in a family member or friend's management of health and/or medications);
  * care recipient must be at least 65 years of age and taking one or more long-term prescription medication;
  * have not participated in this anonymous questionnaire previously

Exclusion Criteria:

* Older adults' exclusion criteria:

  * inability to complete a questionnaire in English.
* Caregivers' exclusion criteria:

  * caregiver's age less than 21 years;
  * caregiver's inability to complete a questionnaire in English.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Potential participants will be selected by convenient sampling from walk-in patients/caregivers who present at the participating pharmacies seeking advice or medication.
Sampling Method: Non-Probability Sample
Enrollment: 1057 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
rPATD questionnaire scorings | up to 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Multi-centres, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No